CLINICAL TRIAL: NCT03199664
Title: Effectiveness of Narrow-band Ultraviolet B Combined With Topical Tacrolimus 0.03% in Treatment of Patients With Vitiligo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Noha Samir, Dermatology resident at South Valley University Students' Hospital, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tcrnbvtlg
Record Dates: First submitted 2017-06-09; First posted 2017-06-27 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (NB-UVB) (Active Comparator): Intervention: patients will be treated with Narrow band ultra violet rays alone for 6 months
  Interventions: Radiation: NB-UVB
- Group B ( combined NB-UVB & Tacrolimus) (Active Comparator): Intervention: patients will be treated with NB-UVB & Tacrolimus 0.03 % ointment for 6 months
  Interventions: Combination Product: NB-UVB & Tacrolimus 0.03%

INTERVENTIONS:
Radiation: NB-UVB — NB-UVB given twice weekly for 6 months
  Arms: Group A (NB-UVB)
Combination Product: NB-UVB & Tacrolimus 0.03% — NB-UVB given twice weekly for 6 months and tacrolimus 0.03 % ointment given for twice daily for the first month of treatment and once daily for the rest 5 months of treatment
  Arms: Group B ( combined NB-UVB & Tacrolimus)

SUMMARY:
The study will compare the effectiveness of combined treatment with NB-UVB and tacrolimus versus NB-UVB alone . Patients will be treated for 6 months and followed up after 3 months .All types of vitiligo will be included except universal vitiligo.

DETAILED DESCRIPTION:
Study approval:

The study will be submitted for approval by the Scientific and Ethical Committees at Faculty of Medicine, South Valley University, Qena. An informed written consent will be obtained from all participants.

Study design:

A randomized controlled trial.

Study population:

The study will include patients who attend the outpatient Clinic of Dermatology, Venereology and Andrology, Faculty of Medicine, South Valley University, with clinical diagnosis of vitiligo. Patients with universal vitiligo, women who are pregnant or lactating at the time of recruitment, children ≤ 2 years old, patients with acute or chronic disease that might affect skin barrier function or patients with history of photosensitivity will be excluded.

Methods:

* Wash out period: ( 4 weeks) During this period, initial medical evaluation will be performed, social demographic data will be collected and patients will be enrolled after obtaining a written consent.
* Test period: (6 months) *Randomization: at the initial visit (visit 0), following the wash out period and before the start of treatment, patients will be randomly assigned to 2 treatment groups; Group (A) : patients will receive NB-UVB sessions twice weekly for 6 months. Initial dose will be 100 mJ/cm2, the dose will be increased by 10% per session.

Group (B) : patients will receive NB-UVB sessions twice weekly for 6 months with the same dose plus topical application of tacrolimus 0.03% ointment twice dialy for the first month of treatment and once dialy for the rest 5 months of treatment.

All Patients will be evaluated before the start of treatment (visit 0) and at monthly intervals for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* all patients with clinical diagnosis of vitiligo.

Exclusion Criteria:

* Patients with universal vitiligo, women who are pregnant or lactating at the time of recruitment, children ≤ 2 years old, patients with acute or chronic disease that might affect skin barrier function or patients with history of photosensitivity.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Vitiligo Area Scoring Index (VASI) | baseline to 9 months
  The percentage of vitiligo involvement is calculated in terms of hand units. One hand unit is approximately equivalent to 1% of the total body surface area. The degree of pigmentation is estimated to the nearest of one of the following percentages: 100% - complete depigmentation, no pigment is present; 90% - specks of pigment present; 75% - depigmented area exceeds the pigmented area; 50% - pigmented and depigmented areas are equal; 25% - pigmented area exceeds depigmented area; and 10% - only specks of depigmentation present. The VASI for each body region is determined by the product of the area of vitiligo in hand units and the extent of depigmentation within each hand unit measured patch.
  Total body VASI = S All body sites [Hand Units] ´ [Residual depigmentation].

SECONDARY OUTCOMES:
Vitiligo Disease Activity (VIDA) score | baseline to 9 months
  The VIDA is a six-point scale for assessing vitiligo activity. Scoring is based on the individual's own opinion of the present disease activity over time. Active vitiligo involves either expansion of existing lesions or appearance of new lesions. Grading is as follows: VIDA Score +4 - Activity of 6 weeks or less duration; +3 - Activity of 6 weeks to 3 months; +2 - Activity of 3 - 6 months;+1 - Activity of 6 - 12 months; 0 - Stable for 1 year or more; and -1 - Stable with spontaneous repigmentation since 1 year or more. A low VIDA score indicates less activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ramdan Saleh, MD, Study Director — Sohag Faculty of Medicine, Sohag university
Locations (1):
- South valley university, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided